CLINICAL TRIAL: NCT00860340
Title: Hemodynamic Effects of Spironolactone in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: xMUO-02
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Hemodynamics; Echocardiographs
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Study patient will take 100mg tablet of Spironolactone
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — 100 mg tablet of Spironolactone (Aldactone) by mouth with half a glass of water.

SUMMARY:
To determine if the beneficial effect of spironolactone in patients with congestive heart failure is in part due to its intrinsic inotropic action.

Randomized, two group placebo controlled, single blind study.

ELIGIBILITY:
Inclusion Criteria:

* CHF
* 21 - 80 years
* Serum creatinine < 2 mg/dL
* Serum potassium 2.7 - 4.5 mg/dL measured within past 4 weeks

Exclusion Criteria:

* Less than 21 years
* Pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-02; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Echocardiogram | 3 measurements 15 minutes apart before drug and 15 minutes for 2 hours after drug
Measure of Kidney function and potassium levels | This will be taken before drug, two hours after and the following day

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Ohio, Toledo, Ohio, United States